CLINICAL TRIAL: NCT04459650
Title: A Pilot Study of the Clinical Effectiveness of Platelet-Rich Plasma (PRP) for the Treatment of Endocrine Therapy-Induced Alopecia (EIA) and Permanent Chemotherapy-Induced Alopecia (pCIA) in Breast Cancer Patients
Brief Title: A Study of PRP Treatment for Hair Loss After Cancer Therapy in Women With Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-133
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Alopecia
Keywords: endocrine therapy induced alopecia; EIA; chemotherapy induced alopecia; pCIA; Memorial Sloan Kettering Cancer Center; 20-133
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Female Breast Cancer Pts (Experimental): Participants include female breast cancer patients who either receive endocrine therapy and suffer from endocrine induced alopecia or suffer from post chemotherapy induced alopecia.
  Interventions: Procedure: Platelet Rich Plasma system

INTERVENTIONS:
Procedure: Platelet Rich Plasma system — Participants will receive PRP obtained with PRP harvesting kits on one side of the scalp and no injections on the other side of the scalp (split-scalp technique). The entire half of the intended scalp will receive inter-follicular injections of PRP under aseptic conditions at the amount of 0.05-0.1 ml/cm2 in a retrograde fashion from deep to superficial, at every centimeter throughout the treated site. For study purposes, Study Day 0 is defined as the first day of injection. Subsequently the patient will continue therapy every 4 weeks for a total of 3 injections (12 weeks).
  Other Names: PRP

SUMMARY:
Participants who enroll in this study will undergo the platelet-rich plasma (PRP) study treatment. Participants will have a sample of blood collected and the platelets will be separated and then injected into half of the participants' scalp every 4 weeks for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age
* Have a clinical diagnosis of endocrine therapy induced alopecia (EIA) for breast cancer:

  * Selective estrogen receptor modulators (tamoxifen, toremifene)
  * Aromatase inhibitors (anastrozole, letrozole, exemestane)
  * Gonadotropin-releasing hormone agonist (leuprolide)

OR

* Must have a clinical diagnosis of chemotherapy induced (pCIA) alopecia with incomplete or absent regrowth of hair > 3 months after completion of chemotherapy without use of endocrine cancer-related therapy (ET) within the last 6 months
* Ludwig stage 1-3 for women
* If patient has a history of use of topical minoxidil and/or systemic spironolactone for alopecia for at least three consecutive months, then a 3 month washout is required prior to start of treatment
* Completed informed consent form

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* History of hair transplantation
* Use of any cosmetic product aimed at improving or correcting the signs of hair loss within 2weeks prior to screening. Note: patients are not permitted to use any hair loss products during the study.
* An active scalp dermatologic condition (e.g. alopecia areata, scalp psoriasis), scalp skin cancer (e.g. BCC, SCC), a pre-existing condition with sequelae on the scalp (e.g. scarring alopecia) or acute infection.
* Hereditary or acquired hematologic/coagulation disorders such as: platelet dysfunction syndrome, critical thrombocytopenia (platelet count <150,000 platelets/ul),hypofibrinogenemia, impaired coagulation, drepanocytosis (sickle cell anemia).
* Actively receiving anticoagulant medication
* Patients taking Aspirin or other NSAIDs such as Nurofen, Voltaren, Diclofenac or Naproxen, or fish-oil supplements because of its anti-platelet activity, can participate, provided medication is interrupted 7 days before beginning of the treatment.
* Planned or previous radiation therapy to the brain
* Vulnerable populations e.g. decisionally impaired (cognitive, psychiatric) or patients who, in the opinion of the investigator have a condition that precludes their ability to provide an informed consent
* Patients taking hair supplements, such as biotin or biosil, can participate, provided hair supplements are washed out 3 months prior to beginning of treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Hair Density | 12 weeks from baseline
  The primary endpoint of this study is the is the relative density in scalp hair at week 12compared to baseline (week 0) between treatment and observation sides of the scalp. The study investigator will use the 7-point GAS (-3 = greatly decreased, -2 = moderately decreased, -1 = slightly decreased, 0 = no change, +1 = slightly increased, +2 = moderately increased, and +3 = greatly increased) to evaluate relative differences in hair density.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony M Rossi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Rossi A, Pan A, Menzer C, Lavin L, Aleissa S, Aleisa A, Alshaikh H, Dranitsaris G, Dusza S, Bravo C, Lacouture ME. Platelet-Rich Plasma Treatment for Endocrine-Induced Alopecia and Persistent Chemotherapy-Induced Alopecia in Breast Cancer Survivors: A Randomized, Controlled, Pilot Study. Dermatol Surg. 2026 Jan 1;52(1):41-47. doi: 10.1097/DSS.0000000000004755. Epub 2025 Jul 8. PMID 40626588
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org